CLINICAL TRIAL: NCT07357220
Title: A Phase Ib/II Clinical Study Evaluating the Safety and Efficacy of AK112 in Combination With VG2025 in Patients With Advanced Colorectal Cancer With Liver Metastases
Brief Title: A Study of AK112 in Combination With VG2025 in Colorectal Cancer With Liver Metastases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Shanghai Virogin Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK112-212
Record Dates: First submitted 2025-12-24; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer With Hepatic Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (VG2025+AK112) (Experimental): VG2025 (Recommended Phase II Dose), Intratumoral Injection, Q4W + AK112 (20mg/kg), ivgtt, Q2W.
  Interventions: Biological: VG2025; Drug: AK112
- Cohort B (AK112) (Experimental): AK112 (20mg/kg), ivgtt, Q2W
  Interventions: Drug: AK112

INTERVENTIONS:
Biological: VG2025 — Recommended Phase II Dose, Intratumoral Injection, Q4W
  Arms: Cohort A (VG2025+AK112)
Drug: AK112 — 20mg/kg, ivgtt, Q2W

SUMMARY:
An open-label, multicenter, phase Ib/II study of AK112 in combination with VG2025 for advanced colorectal cancer with liver metastases.

DETAILED DESCRIPTION:
This open-label, multicenter, phase Ib/II clinical study aims to evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of AK112 in combination with VG2025, in the treatment of advanced colorectal cancer with liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age≥18 years and ≤ 75 years
3. Histologically or cytologically confirmed unresectable colorectal cancer with liver metastases; adenocarcinoma type
4. Disease progression after first- or second-line standard therapy
5. At least one measurable disease based on RECIST v1.1
6. ECOG status of 0 or 1
7. Estimated life expectancy≥3 months
8. Adequate organ function
9. Patients with fertility are willing to use an adequate method of contraception

Exclusion Criteria:

1. Histologically or cytologically confirmed non-adenocarcinoma or mixed-type tumors with adenocarcinoma component ≤70%
2. Known dMMR or MSI-H
3. Known RAS or BRAF mutations
4. Participation in another clinical trial
5. Systemic anticancer therapy within 4 weeks, small molecule therapy within 2 weeks, antitumor traditional Chinese medicine within 2 weeks before first dose
6. Prior immunotherapy other than anti-PD-(L)1 agents
7. Live attenuated vaccine within 28 days before or during study treatment and 90 days after last dose
8. Active malignancy within the past 3 years
9. Known spinal cord compression, active brain or leptomeningeal metastases.
10. Significant bleeding events requiring transfusion, invasive intervention, or hospitalization within 3 months before first dose
11. Serious infection within 28 days, or systemic anti-infective therapy within 14 days before first dose (except antiviral therapy for hepatitis B/C)
12. Active herpesvirus infection with clinical manifestations
13. Active autoimmune disease
14. Known immunodeficiency
15. Known allergy to study drug or excipients, or history of severe allergic reactions to other vaccines
16. History of allogeneic organ or hematopoietic stem cell transplantation.
17. Clinically significant liver disease
18. Any other situations that are not suitable for inclusion in this study judged by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities (DLTs) | From Day 1 to Day 28 after the first tumour vaccine was administrated in safety run-in cohorts
  Number of participants who meet the criteria of dose-limiting toxicities (DLTs) in DLT observation period
Number of participants with adverse events (AEs) and severity | From ICF up to 30 days after last study treatment
  Number of participants experiencing adverse events (AEs) and severity, graded according to CTCAE v5.0
Objective Response Rate (ORR) | Time Frame: Up to 2 years
  Proportion of participants with complete response (CR) or partial response (PR), as assessed by RECIST version 1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 years
  Time from the date of enrollment until the first documentation of disease progression or death due to any cause, whichever occurs first, as assessed by RECIST version 1.1
Disease control rate (DCR) | Up to 2 years
  Proportion of participants with complete response (CR), partial response (PR), or stable disease (SD), as assessed by RECIST version 1.1
Duration of response (DoR) | Up to 2 years
  Time from the first documentation of objective response to the first documented disease progression as assessed by RECIST version 1.1 or death due to any cause, whichever occurs first
Time to response (TTR) | Up to 2 years
  Time from the start of the treatment to the first objective tumor response observed for patients who achieved complete response (CR) or partial response (PR), as assessed by RECIST version 1.1
Overall survival (OS) | Up to 2 years
  Time from the date of enrollment to death from any cause
Observed concentrations of AK112 | Up to 2 years
  Observed serum concentrations of AK112 at different time points after AK112 administration
Number of participants with detectable anti-drug antibodies (ADAs) to AK112 | Up to 2 years
  Number of participants who develop detectable anti-drug antibodies (ADAs) to AK112

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine，No. 79, Qingchun Road, Shangcheng District, Hangzhou City, Zhejiang Province, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No